CLINICAL TRIAL: NCT04978090
Title: Pilot Study Evaluating the Safety and Efficacy of a Patient-Specific Enteroatmospheric Fistula Isolation and Management Device Independent of Negative Pressure Wound Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Bernard (Other)
Responsible Party: Sponsor-Investigator, Andrew Bernard, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 46641
Record Dates: First submitted 2021-07-01; First posted 2021-07-27 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Fistula; Abdominal Injury; Negative Pressure Wound Therapy
Keywords: Open abdominal; Wound care
MeSH Terms: conditions — Fistula; Abdominal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Enteroatmospheric fistula (EAF) management solution (Experimental): Participants will receive a custom fitted device designed to isolate EAF effluent independent of negative pressure wound therapy (NPWT) utilizing 3D printing technology to design a participant-matched device that more easily and effectively separates the participant's fistula and any emanated intestinal contents surrounding the wound.
  Interventions: Device: 3D printed EAF management device

INTERVENTIONS:
Device: 3D printed EAF management device — Participants will receive a customized 3D printed device based on the EAF's output, size, shape, location, depth, and the participant's wound bed.

SUMMARY:
This study aims to assess the efficacy of a custom fitted device designed to isolate enteroatmospheric fistulas effluent independent of negative pressure wound therapy and to evaluate the effects on the device related to dressing changes, time required for dressing changes, management costs, and the ease of use.

ELIGIBILITY:
Inclusion Criteria:

* Stable condition, as determined by attending physician
* Has enteroatmospheric fistula (EAF) in the setting of open abdomen
* EAF is determined to require surgical resolution

Exclusion Criteria:

* Unstable condition, as determined by attending physician
* Significant risk of complication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bernard, MD, FACS, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Started | 2
Completed | 0
Not Completed | 2
Not completed — unable to adequately fit device | 2

BASELINE CHARACTERISTICS:
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Inpatient Participant Pain Rating
Description: Participants will be asked to rate their pain on a scale of 1-10, where 10 indicates more pain.
Time Frame: Daily from admission to discharge, up to 1 year
Population: Two participants were enrolled in this study. Due to the possibility that the participants could reasonably be identified due to low enrollment, data cannot be presented.
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Outpatient Participant Pain Rating
Description: Participants will be asked to rate their pain on a scale of 1-10, where 10 indicates more pain.
Time Frame: Weekly from discharge until fistula resolves or study ends, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

3. Primary Outcome: Change in Inpatient Participant Mobility Assessment
Description: Mobility will be assessed by asking the participant to select the following statement that most accurately describes their mobility: a. completely immobile; b. unable to sit up supported for less than 10 minutes; c. able to sit supported for more than 10 minutes; d. able to sit unsupported, can lift arms; e. can stand up and pivot torso; or f. can walk and move with minimal assistance required.
Time Frame: Daily from admission to discharge, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

4. Primary Outcome: Change in Outpatient Participant Mobility Assessment
Description: as for outcome 3
Time Frame: Weekly from until fistula resolves or study ends, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

5. Primary Outcome: Change in Number of Required Wound Dressing Changes - Inpatient
Description: The number of dressing changes will be tracked for inpatients on a daily bases.
Time Frame: Daily from admission to discharge, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

6. Primary Outcome: Change in Number of Required Wound Dressing Changes - Outpatient
Description: The number of dressing changes will be tracked for outpatients on a daily bases.
Time Frame: Daily from discharge until fistula resolves or study ends, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

7. Primary Outcome: Change in Perceived Usefulness - Inpatient
Description: Inpatient participants will be asked three questions about the perceived usefulness of the device. The questions use a 5-point Likert scale ranging from strongly disagree to strongly agree, where strongly agree indicates a higher perceived usefulness.
Time Frame: Daily from admission to discharge, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

8. Primary Outcome: Change in Perceived Usefulness - Outpatient
Description: Outpatient participants will be asked two questions about the perceived usefulness of the device. The questions use a 5-point Likert scale ranging from strongly disagree to strongly agree, where strongly agree indicates a higher perceived usefulness.
Time Frame: Weekly from discharge until fistula resolves or study ends, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

9. Primary Outcome: Change in Perceived Ease of Use - Inpatient
Description: Inpatient participants will be asked four questions about the perceived ease of use of the device. The question uses a 5 point Likert scale ranging from strongly disagree to strongly agree, where strongly agree indicates a higher perceived ease of use.
Time Frame: Daily from admission to discharge, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

10. Primary Outcome: Change in Perceived Ease of Use - Outpatient
Description: as for outcome 9
Time Frame: Weekly from discharge until fistula resolves or study ends, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

11. Primary Outcome: Change in Average Time of Required Fistula-specific Dressing Changes - Inpatient
Description: The time required to change the wound dressings will be recorded.
Time Frame: Daily from admission to discharge, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

12. Secondary Outcome: Infection Rates
Description: The number of infections in participants that are related to the device will be recorded.
Time Frame: Through duration of study, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Observed Leakages
Description: The number of observed leakages in participants that are related to the device will be recorded.
Time Frame: Through duration of study, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

14. Secondary Outcome: Length of Stay
Description: Length of stay in hospital
Time Frame: Through duration of study, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

15. Secondary Outcome: Fistula Resolution Time
Description: Fistula resolution time for participants
Time Frame: Through duration of study, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

16. Secondary Outcome: Complication Occurrences
Description: The number of complication occurrences related to the device will be recorded.
Time Frame: Through duration of study, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

17. Other Pre Specified Outcome: Cost Analysis of the 3D Printed Device
Description: The cost of the patient management with the device will be estimated
Time Frame: Weekly from beginning of study until the end of the study, up to 1 year
Population: as for outcome 1
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Two participants were enrolled in this study. Due to the possibility that the participants could reasonably be identified due to low enrollment, data cannot be presented.
Description: Two participants were enrolled in this study. Due to the possibility that the participants could reasonably be identified due to low enrollment, data cannot be presented.
Arm/Group | Enteroatmospheric Fistula (EAF) Management Solution
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT04978090/Prot_ICF_000.pdf